CLINICAL TRIAL: NCT04582448
Title: A Trial Investigating the Pharmacokinetic Properties of Insulin Icodec After Administration in Different Injection Regions in Subjects With Type 2 Diabetes
Brief Title: A Study Looking at How Insulin Icodec is Taken up in the Blood When Administered in Different Injection Sites in People With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4572; U1111-1244-4495 (Other: World Health Organization (WHO)); 2019-004660-21 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-10-08; First posted 2020-10-09 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Insulin icodec treatment sequence with injection region abdomen (Experimental): Each subject will be randomised to one of six treatment sequences, consisting of three single-dose administrations of insulin icodec (s.c. in the abdomen, the upper arm and the thigh) in a balanced manner on three separate treatment visits.
  Interventions: Drug: Insulin icodec
- Insulin icodec treatment sequence with injection region upper arm (Experimental): Each subject will be randomised to one of six treatment sequences, consisting of three single-dose administrations of insulin icodec (s.c. in the abdomen, the upper arm and the thigh) in a balanced manner on three separate treatment visits.
  Interventions: Drug: Insulin icodec
- Insulin icodec treatment sequence with injection region thigh (Experimental): Each subject will be randomised to one of six treatment sequences, consisting of three single-dose administrations of insulin icodec (s.c. in the abdomen, the upper arm and the thigh) in a balanced manner on three separate treatment visits.
  Interventions: Drug: Insulin icodec

INTERVENTIONS:
Drug: Insulin icodec — A single dose of insulin icodec administered subcutaneously (s.c. - under the skin) Injection in the belly, upper arm and thigh on different occasions.

SUMMARY:
This study is comparing the concentration of a single dose of insulin icodec when administered in the belly, upper arm and thigh on different occasions.

Participants will receive one injection of insulin icodec on three different occasions, each time injected at a different site, i.e. either on our belly, upper arm or thigh.

The study will last for about 34 weeks. Participants will have 23 visits with the study doctor. Informed Consent (V0) visit and screening visit (V1) will be performed on two different days. The informed consent visit may be performed via telephone to minimize personal contact with site staff during the coronavirus outbreak.

Women cannot take part if pregnant, breast- feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-69 years (both inclusive) at the time of signing informed consent
* Body mass index between 18.5 and 38.0 kg/m^2 (both inclusive)
* Diagnosed with type 2 diabetes mellitus above or equal to 180 days prior to the day of screening
* HbA1c (glycated haemoglobin) below or equal to 9.0 percentage at screening
* Current daily basal insulin treatment of 0.2-1.0 (I)U/kg/day (both inclusive) with or without any of the following anti-diabetic drugs/regimens with stable doses above or equal to 90 days prior to the day of screening:
* Any metformin formulation
* Other oral antidiabetic drugs: DPP-4 inhibitors / SGLT2 inhibitors / Oral combination products (for the allowed individual oral antidiabetic drugs)
* Oral or injectable GLP-1 (glucagon-like peptide 1) Receptor Agonists

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
AUCIco,0-inf,SD, Area under the serum insulin icodec concentration-time curve after a single dose | Day 1
  From 0 hours until infinity after trial product administration (pmol*h/L)

SECONDARY OUTCOMES:
Cmax,Ico,SD, Maximum observed serum insulin icodec concentration after a single dose | Day 1
  From 0 hours until infinity after trial product administration (pmol/L)
tmax,Ico,SD, Time to maximum observed serum insulin icodec concentration after a single dose | Day 1
  From 0 hours until infinity after trial product administration (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Plum-Morschel L, Andersen LR, Hansen S, Hovelmann U, Krawietz P, Kristensen NR, Lehrskov LL, Haahr H. Pharmacokinetic and Pharmacodynamic Characteristics of Insulin Icodec After Subcutaneous Administration in the Thigh, Abdomen or Upper Arm in Individuals with Type 2 Diabetes Mellitus. Clin Drug Investig. 2023 Feb;43(2):119-127. doi: 10.1007/s40261-022-01243-6. Epub 2023 Jan 11. PMID 36631720